CLINICAL TRIAL: NCT03698708
Title: Longitudinal Test of Adherence & Control in Kids New to Type 1 Diabetes & 5-9 Years Old
Brief Title: Cognitive Adaptations to Reduce Emotional Stress Associated With Type 1 Diabetes
Acronym: CARES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01DK100779-05 (NIH)
Record Dates: First submitted 2018-10-03; First posted 2018-10-09 (Actual); Results first posted 2022-02-11 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-01

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CARES Intervention- 12 sessions (Experimental): Participants in the intervention will participate in 12 weekly group-based telemedicine intervention sessions (up to 60 minutes each) with other parents/caregivers of children with T1D. Intervention sessions focus on cognitive-behavioral therapy to treat depression, including identifying cognitive distortions, cognitive restructuring, behavioral activation, coping strategies, and learning diabetes management skills.
  Interventions: Behavioral: CARES Intervention
- CARES Intervention- 8 sessions (Experimental): Participants in the intervention will participate in 8 weekly group-based telemedicine intervention sessions (up to 60 minutes each) with other parents/caregivers of children with T1D. Intervention sessions focus on cognitive-behavioral therapy to treat depression, including identifying cognitive distortions, cognitive restructuring, behavioral activation, coping strategies, and learning diabetes management skills.
  Interventions: Behavioral: CARES Intervention

INTERVENTIONS:
Behavioral: CARES Intervention — A group-based telemedicine intervention to treat depression in parents/caregivers of children with T1D using a cognitive-behavioral approach.

SUMMARY:
The purpose of this study is to evaluate a new intervention (CARES: Cognitive Adaptations to Reduce Emotional Stress Associated with Type 1 Diabetes) designed to reduce caregiver depressive symptoms in families of children with T1D. This is a pilot in which all enrolled parents/caregivers will be placed in the intervention group to assess initial pre- to post-treatment impact of the intervention on parent/caregiver depression, distress, and diabetes-related outcomes (e.g., glycemic control).

ELIGIBILITY:
Inclusion Criteria:

* Parent/primary caregiver of a child diagnosed with T1D between 5-12 years old
* Parent/caregiver elevated depression symptoms on the CESD-R (score ≥ 16 at time of screening)
* Child with T1D receiving intensive insulin regimen by multiple dose injections (MDI) or continuous subcutaneous insulin infusion (pump)

Exclusion Criteria:

* Child with T1D currently in foster care or not living with legal guardian
* Child with evidence of type 2 diabetes or monogenic diabetes
* Child with a co-morbid chronic illness (e.g., renal disease) that requires ongoing care beyond T1D
* Children who are chronically using medications that may impact glycemic control (i.e., systemic steroids)
* Parents/caregivers who do not speak English (currently there is no way to recruit non-English speaking families because the study questionnaires are only available in English)

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 37 (Actual)
Dates: Start 2019-01-20 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Children's Mercy Hospital, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Case H, Williams DD, Majidi S, Ferro D, Clements MA, Patton SR. Longitudinal associations between family conflict, parent engagement, and metabolic control in children with recent-onset type 1 diabetes. BMJ Open Diabetes Res Care. 2021 Oct;9(1):e002461. doi: 10.1136/bmjdrc-2021-002461. PMID 34645616
- [Derived] McConville A, Noser AE, Nelson EL, Clements MA, Majidi S, Patton SR. Depression as a predictor of hypoglycemia worry in parents of youth with recent-onset type 1 diabetes. Pediatr Diabetes. 2020 Aug;21(5):909-916. doi: 10.1111/pedi.13039. Epub 2020 May 29. PMID 32410305

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruited in clinic, by telephone, and through email
Pre-assignment Details: The study recruited parents/caregivers as participants only. Parents gave permission for researchers to collect an HbA1c level for their child. Children did not participate in the treatment.
Period: Overall Study
Arm/Group | CARES Intervention- 12 Sessions | CARES Intervention- 8 Sessions
Started | 17 | 20
Completed | 13 | 16
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Population: Primary outcomes were parent report variables: diabetes distress, depressive symptoms, fear of hypoglycemia, treatment satisfaction. As an exploratory variable, we examined children's HbA1c level.
Groups:
- Total: Total of all reporting groups
Arm/Group | CARES Intervention- 12 Sessions | CARES Intervention- 8 Sessions | Total
Number analyzed (Participants) | 17 | 20 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 20 | 37
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.29 (7.49) | 38.25 (6.07) | 39.65 (6.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 20 | 36
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 16 | 19 | 35
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 15 | 16 | 31
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 0 | 1 | 1
Problem Areas in Diabetes-PR [Mean (Standard Deviation); unit: units on a scale] — This is a validated measure of diabetes distress. Parents/Caregivers completed this measure. Higher scores reflect more distress. Range 0-72.
  units on a scale | 32.65 (11.87) | 39.69 (14.72) | 36.45 (13.77)
Center for Epidemiological Study Depression Scale Revised [Mean (Standard Deviation); unit: units on a scale] — This is a measure of depressive symptoms. Parents/Caregivers completed this measure. Higher scores reflect more depressive symptoms. Score range 0-60.
  units on a scale | 16.12 (11.21) | 11.25 (11.08) | 13.49 (10.17)
Hypoglycemia Fear Survey-Parents [Mean (Standard Deviation); unit: units on a scale] — This is a measure of hypoglycemia fear. Parents/Caregivers completed this measure. Higher scores reflect greater fear of hypoglycemia. Scores range 25-125.
  units on a scale | 66.47 (14.12) | 67.95 (16.27) | 67.27 (15.13)

OUTCOME MEASURES:

1. Primary Outcome: Problem Areas in Diabetes Survey - Parent Revised (PAID-PR)
Description: Problem Areas in Diabetes Survey - Parent Revised (PAID-PR); Parents' perceptions of diabetes-related distress, which can encompass fear, sadness, grief, anger, burn-out, and guilt. Higher scores reflect greater perceived distress (range: 0-72)
Time Frame: absolute value Post-treatment (week 24)
Population: reflects sample of parents who completed the treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CARES Intervention- 12 Sessions | CARES Intervention- 8 Sessions
Number analyzed (Participants) | 13 | 16
units on a scale | 32.65 (11.87) | 39.69 (14.72)
Statistical Analysis 1: Comparison: CARES Intervention- 12 Sessions vs CARES Intervention- 8 Sessions; Test type: Superiority; repeated measures ANOVA; cohen's d = .88

2. Primary Outcome: Center for Epidemiologic Studies - Depression Scale Revised (CESD-R)
Description: Center for Epidemiologic Studies - Depression Scale Revised (CESD-R); measure of parental depressive symptoms. Used as a secondary marker of improvement. Higher scores reflect greater occurrence of depressive symptoms (range: 0-60)
Time Frame: absolute value at Post-treatment (week 24)
Population: data for parents who completed treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CARES Intervention- 12 Sessions | CARES Intervention- 8 Sessions
Number analyzed (Participants) | 13 | 16
units on a scale | 15.85 (11.15) | 12.12 (9.24)
Statistical Analysis 1: Comparison: CARES Intervention- 12 Sessions vs CARES Intervention- 8 Sessions; Test type: Superiority; repeated measures ANOVA; cohen's d = .22

3. Secondary Outcome: Hypoglycemia Fear Survey (HFS-P)
Description: Hypoglycemia Fear Survey (HFS-P); measure of parents fear of hypoglycemia, a secondary symptom that can relate to distress; Higher scores reflect greater perceptions of fear as well as use of hypoglycemia avoidance behaviors (range: 25-125).
Time Frame: absolute value Post-treatment (week 24)
Population: reflects data from parents who completed treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CARES Intervention- 12 Sessions | CARES Intervention- 8 Sessions
Number analyzed (Participants) | 13 | 16
units on a scale | 61.92 (12.23) | 63.56 (13.36)
Statistical Analysis 1: Comparison: CARES Intervention- 12 Sessions vs CARES Intervention- 8 Sessions; Test type: Superiority; repeated measures ANOVA; cohen's d = .05

4. Secondary Outcome: Diabetes Family Conflict Scale (DFCS)
Description: Diabetes Family Conflict Scale (DFCS): parents perceptions of diabetes-related family conflict. Higher scores reflect greater perceived conflict, which includes arguing about daily diabetes tasks and periodic diabetes tasks (range= 19-57)
Time Frame: absolute value Post-treatment (week 24)
Population: reflects data for parents who completed treatment only
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CARES Intervention- 12 Sessions | CARES Intervention- 8 Sessions
Number analyzed (Participants) | 13 | 16
units on a scale | 23.0 (2.64) | 25.62 (7.34)
Statistical Analysis 1: Comparison: CARES Intervention- 12 Sessions vs CARES Intervention- 8 Sessions; Test type: Superiority; repeated measures ANOVA; cohen's d = .14

5. Secondary Outcome: Hemoglobin A1c (HbA1c)
Description: Proxy measure of glycemic control over the past 12 weeks
Time Frame: absolute value at Post-treatment (week 24)
Population: reflects data for children of parents who completed treatment only
Measure: Mean (Standard Deviation); unit: percentage of glycated hemoglobin cells
Arm/Group | CARES Intervention- 12 Sessions | CARES Intervention- 8 Sessions
Number analyzed (Participants) | 13 | 16
percentage of glycated hemoglobin cells | 8.13 (0.88) | 8.45 (1.64)
Statistical Analysis 1: Comparison: CARES Intervention- 12 Sessions vs CARES Intervention- 8 Sessions; Test type: Superiority; repeated measures ANOVA; cohen's d = .09

6. Other Pre Specified Outcome: Treatment Satisfaction Survey
Description: Treatment Satisfaction Survey; Intervention acceptability and satisfaction. This measure was designed for this pilot study. Higher scores reflect greater satisfaction/acceptability (range: 15-75).
Time Frame: absolute value at post-treatment (week 12)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CARES Intervention- 12 Sessions | CARES Intervention- 8 Sessions
Number analyzed (Participants) | 13 | 16
score on a scale | 53.93 (5.77) | 49.76 (9.44)
Statistical Analysis 1: Comparison: CARES Intervention- 12 Sessions vs CARES Intervention- 8 Sessions; Test type: Superiority; ANOVA; Mean Difference (Final Values) = -4.16, 95% CI 2-sided [-10.07 to 1.74]

ADVERSE EVENTS:
Time Frame: through study completion, average 7 months
Description: Behavioral trial; deemed less than minimum risk by the IRB of record
Groups:
- CARES Intervention- 12 Sessions: Participants in the intervention will participate in 12 weekly group-based telemedicine intervention sessions (up to 60 minutes each) with other parents/caregivers of children with T1D. Intervention sessions focus on cognitive-behavioral therapy to treat depression, including identifying cognitive distortions, cognitive restructuring, behavioral activation, coping strategies, and learning diabetes management skills.
  CARES Intervention: A group-based telemedicine intervention to treat depression in parents/caregivers of children with T1D using a cognitive-behavioral approach.
  Children did not receive treatment and were not monitored for adverse events.
- CARES Intervention- 8 Sessions: Participants in the intervention will participate in 8 weekly group-based telemedicine intervention sessions (up to 60 minutes each) with other parents/caregivers of children with T1D. Intervention sessions focus on cognitive-behavioral therapy to treat depression, including identifying cognitive distortions, cognitive restructuring, behavioral activation, coping strategies, and learning diabetes management skills.
  CARES Intervention: A group-based telemedicine intervention to treat depression in parents/caregivers of children with T1D using a cognitive-behavioral approach.
  Children did not receive treatment and were not monitored for adverse events.
Arm/Group | CARES Intervention- 12 Sessions | CARES Intervention- 8 Sessions
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/20
Other Adverse Events (participants affected / at risk) | 0/17 | 0/20

LIMITATIONS AND CAVEATS:
Original proposal called to pilot the CARES in n=12; we recruited additional participants to simultaneously trial the 8-session CARES version. These results are preliminary and require confirmation in a fully powered comparative effectiveness trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-04): https://cdn.clinicaltrials.gov/large-docs/08/NCT03698708/Prot_SAP_000.pdf